CLINICAL TRIAL: NCT07212504
Title: Effect of Accelerated Neuromodulation of Anterior Cingulate Cortex to Enhance Cognition in Older Adults With Mild Memory Problems
Acronym: NACC-EC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rotman Research Institute at Baycrest (Other)
Responsible Party: Principal Investigator, Linda Mah, MD, Clinician Scientist, Rotman Research Institute at Baycrest
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-04
Record Dates: First submitted 2025-09-11; First posted 2025-10-08 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment (MCI); Subjective Cognitive Decline (SCD)
Keywords: Mild Cognitive Impairment; Subjective Cognitive Decline; Transcranial Magnetic Stimulation (TMS); Intermittent Theta Burst Stimulation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 20-40 sessions of iTBS dTMS and 6-weeks of online cognitive remediation (Experimental)
  Interventions: Device: Active Brainsway H7-Coil Deep TMS System
- 20-40 sessions of sham stimulation and 6-weeks of online cognitive remediation (Sham Comparator)
  Interventions: Device: Sham Brainsway H1-Coil Deep TMS System

INTERVENTIONS:
Device: Active Brainsway H7-Coil Deep TMS System — Deep Transcranial Magnetic Stimulation (dTMS) is a new form of TMS which allows direct stimulation of deeper neuronal pathways than the standard TMS. The H-coil is a novel dTMS coil designed to allow deeper brain stimulation without a significant increase of electric fields induced in superficial cortical regions. dTMS will be administered 6-8 times a day for 2-5 consecutive days.
  Arms: 20-40 sessions of iTBS dTMS and 6-weeks of online cognitive remediation
Device: Sham Brainsway H1-Coil Deep TMS System — In addition to the active H7-coil, a sham coil is included in the H1-coil helmet.The sham treatment will be administered using the H1-coil helmet 6-8 times a day for 2-5 consecutive days.
  Arms: 20-40 sessions of sham stimulation and 6-weeks of online cognitive remediation

SUMMARY:
The goal of this clinical trial is to test whether an accelerated deep Transcranial Magnetic Stimulation (dTMS) protocol in combination with cognitive training can improve cognitive abilities in older adults with Subjective Cognitive Decline (SCD) or Mild Cognitive Impairment (MCI). The study will look at whether it is safe and tolerable to use accelerated dTMS to enhance the benefits of cognitive training in older adults, and will also gather early information on the effects of accelerated dTMS on memory and other cognitive abilities.

DETAILED DESCRIPTION:
This study will examine the effects of combining cognitive remediation with accelerated intermittent theta burst stimulation (a-iTBS) using the H7 deep Transcranial Magnetic Stimulation (dTMS) coil to target the anterior cingulate cortex (ACC) in older adults aged 55-85 with MCI or SCD. Thirty older adults will participate in a single site, double-blind, randomized sham-controlled trial using an accelerated schedule of multiple dTMS sessions per day for 2-5 consecutive days, followed by 6 weeks of online cognitive remediation for both sham and dTMS interventions. The primary goal of the study is to establish the feasibility of an a-iTBS protocol combined with cognitive training in older adults with Mild Cognitive Impairment (MCI) and Subjective Cognitive Decline (SCD) and to obtain preliminary evidence of treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 55 - 85 years of age (on the day of randomization)
* are male or post-menopausal female
* have a diagnosis of mild cognitive impairment (MCI) based on Montreal Cognitive Assessment score < 26 or where available, results from clinical neuropsychological assessment, OR subjective memory concerns and first degree relative, living or deceased, with a probable or confirmed diagnosis of AD
* score 24 or higher on the Mini Mental State Examination (MMSE)
* are willing to provide informed consent
* are able to follow the treatment schedule
* are stable on medications for 2 months and are not expected to change medication during the entire study period (if they are taking medications)
* have a satisfactory safety screening questionnaire for TMS

Exclusion Criteria:

* have a metal plate in their head(such as an ear implant, implanted brain stimulators, aneurysm clips). Dental devices and implants that are non-magnetic are safe.
* have known increased pressure or a history of increased pressure in their brain, which may increase their risk for having seizures
* have a cardiac pacemaker
* have an implanted medication pump
* have a central venous line
* have a history of any psychotic disorder, bipolar disorder, eating disorder, obsessive compulsive disorder, post-traumatic stress disorder, or dementia
* have a history of substance abuse in the last 6 months
* have a history of stroke or other brain lesions
* have a personal history of epilepsy
* have a family history of epilepsy
* are a pregnant or breast-feeding woman
* have a history of abnormal MRI of the brain
* have untreated hypo- or hyper-thyroidism
* have unstable medical condition(s)
* have any other known contraindications to TMS
* are on unstable doses of any psychotropic medication such as antidepressants, antipsychotic, mood stabilizers or memory enhancing medications
* regularly use benzodiazepines or other hypnotics within 2 weeks of randomization

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of dTMS sessions attended by participants | 1 week
Incidence and type of of adverse events experienced during treatment (participant-reported tolerability) based on the Adverse Events Questionnaire (AEQ) | 9 weeks
  The AEQ asks about symptoms related immediately after TMS administration where patients rate symptom severity from 1 (absent) to 4 (severe) and whether they believe it is related to TMS from 1 (no) to 5 (definitely).
The number of participants who prematurely withdraw and reasons for withdrawal | 9 weeks
Change from baseline memory scores on computerized neuropsychological battery following the final session on day 5 | 9 weeks
  Memory score from memory tests in the neuropsychological battery at baseline will be compared to after 5 days of TMS and after 6 weeks of cognitive training the active intervention group compared to the sham. A higher memory score indicates better memory performance. An effect size (Cohen's d) of 0.5 will be considered a minimally important effect size.
Change from baseline executive function scores on computerized neuropsychological battery following final session on day 5 | 9 weeks
  Executive function scores from tests on the neuropsychological battery will be compared from baseline to after days of dTMS and after 6 weeks of cognitive training in the active intervention group compared to sham. A higher score on these tests indicate greater executive functioning. An effect size (Cohen's d) of 0.5 will be considered a minimally important effect size.

SECONDARY OUTCOMES:
The change in baseline in scores on the Geriatric Anxiety Inventory (GAI) following 5 days of dTMS | 1 week
  The GAI is a 20-item self-report measure of anxiety developed for older adults. Administration time is approximately 5 minutes. The GAI scores range from 0-20, with higher scores indicating more anxiety.
The change in resting state activity as measured with electroencephalography (EEG) following 5 days of dTMS | 1 week
The change in slow wave activity in the posterior default mode network (posterior cingulate cortex) as measured with MEG following 5 days of dTMS | 1 week
The change in functional connectivity within the default mode network based on Magnetic Resonance Imaging (MRI) following 5 days of dTMS | 1 week
The change in baseline in scores on the Geriatric Depression Scale (GDS) | 1 week
  GDS is a 15-item self-report scale that measures an elderly individual's mood. A score greater than 5 suggests that the individual may be depressed. Administration time is approximately 5 minutes. GDS scores range from 0-15 with a greater score indicating greater depressive symptoms.
The change in baseline slow wave as measured with electroencephalography (EEG) following 5 days of dTMS | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Linda Mah, MD, Principal Investigator — Baycrest Rotman Research Institute
Locations (1):
- Rotman Research Institute at Baycrest, Toronto, Ontario, Canada